CLINICAL TRIAL: NCT04459182
Title: Circulating Exosomes and Endothelial Dysfunction in Patients With Obstructive Sleep Apneas Hypopneas Syndrome(OSA): EXODYS
Brief Title: Circulating Exosomes and Endothelial Dysfunction in Patients With Obstructive Sleep Apneas Hypopneas Syndrome
Acronym: EXODYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-A01855-34
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Endothelial Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endothelial dysfunction (DE+) (Active Comparator): obsese patient with OSA (AHI>15) and endothelial dysfunction
  Interventions: Diagnostic Test: ENDOPAT
- No endothelial dysfunction (DE-) (Sham Comparator): obsese patient with OSA (AHI>15) and no endothelial dysfunction
  Interventions: Diagnostic Test: ENDOPAT

INTERVENTIONS:
Diagnostic Test: ENDOPAT — digital plethysmography

SUMMARY:
Evaluation of miRNA contained in exosomes in obese and OSA patients with endothelial dysfunction evaluated by digital plethysmography (ENDOPAT) compared to obese and OSA patients without endothelial dysfunction.

DETAILED DESCRIPTION:
The aim of the study is to compare the content of exosomes between two goups of 20 patients, with and without endothelial dysfucntion.

the endothelial function will be evaluated after polysomnography, on obese patients with OSA (AHI >15).

ELIGIBILITY:
Inclusion Criteria:

* adult subject
* Subject understands the study protocol and is willing and able to comply with study requirements and sign informed consent
* Subject with OSA (defined by AHI >15/h)

Exclusion Criteria:

* cardiac or vascular desease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
miRNA cointained in exosomes | immediately after the consultation
  compare exosome content between obese-OSA patients with endothelial dysfunction and without

CONTACTS AND LOCATIONS:
Overall Officials: GAGNADOUX Frédéric, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- Frédéric GAGNADOUX, Angers, France

IPD SHARING:
Plan to Share IPD: No